CLINICAL TRIAL: NCT05697458
Title: Evaluation and Prognostic Value of Iliac Arterial Calcifications Determined With Computerized Tomography and Bone Remodeling Biomarkers in Patients With Kidney Transplantation
Brief Title: Vascular Calcifications in Kidney Transplant Recipient
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Sponsor
Other Study IDs: 3105
Record Dates: First submitted 2022-12-26; First posted 2023-01-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Arterial Calcification; Kidney Failure; Kidney Transplant; Complications
Keywords: kidney transplantation; end stage renal disease; arterial calcifications
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: In kidney transplant recipients the investigators will perform pretransplant computerized tomography for assessment of iliac arteries calcifications.
  From their blood, the bone remodeling biomarkers will be determined in the perioperative period.
  The one year patient and graft survival will be determined for included patients.
  Interventions: Other: computerized tomography scanning

INTERVENTIONS:
Other: computerized tomography scanning — In all patients the investigators will perform CT for determination of iliac arteries calcifications

SUMMARY:
Kidney transplant candidates undergo extensive diagnostic evaluation aimed at assessing their cardiovascular (CV) risk, which remains the leading cause of disability and death in this patient population. This includes among others an assessment of the iliac arterial calcification. Chronic kidney disease (CKD) patients have an increased incidence of arterial calcifications due to many factors, such as increased age, hyperparathyroidism, diabetes mellitus and hypercholesterolemia. Furthermore, the severity of pelvic arterial calcifications may impact the surgical planning of kidney transplantation (KT), choice of anastomosis site, complexity of the surgery, and patient and graft survival. Vascular calcifications are recognized as a good biomarker of overall cardiovascular burden. Although computerized tomography (CT) is the imaging modality of choice for calcification evaluation, compared to pelvic X-ray and Doppler ultrasound, it is not officially included in the guidelines of different international associations, which offer general recommendations for the assessment of iliac vessels. Nevertheless, centers are increasingly using CT in their pretransplant workup, either routinely or only in patients with increased CV risk. Also, impaired bone metabolism and its consequences have an important role in the development of vascular calcification.

The investigators will determine the relationship between calcification burden of iliac arteries which will be assessed on CT and the serum level of bone remodeling biomarkers, including parathyroid hormone, (PTH), calcium, phosphates, OPG/RANK/RANKL (engl. osteoprotegerin/receptor activator of nuclear factor (NF)-κΒ/RANK ligand) and Gla-Rich protein (GLP). According to investigator knowledge, this will be the first prospective study that will correlate the degree of iliac arteries calcification based on CT analyses with the serum level of various bone remodeling markers, and their impact on clinical outcome in kidney transplant recipients.

The investigators expect this research to improve insights into incidence and distribution of iliac artery calcifications in patients following kidney transplantation, their correlation with clinical data and bone remodeling markers and confirm the appropriateness of using computerized tomography in a routine pretransplantation work-up.

DETAILED DESCRIPTION:
The hypothesis of this study is that incidence and severity of arterial calcification raise with age of the patient and time spent on hemodialysis. Additionally, poorer graft and patient survival and overall risk for future cardiovascular events correlate with the severity of arterial calcifications following successful kidney transplantation.

Study will include 50 patients who will undergo kidney transplantation. Non-contrast CT scan of abdomen and pelvis will be performed, and blood level of bone remodeling markers will be determined in all patients.

Two radiologists will independently assess the severity of iliac artery calcifications, by using quantitative scoring system developed by Davis et al. and newly developed pelvic calcification score.

Pelvic calcification score (PCS) will be determined by assessing common iliac artery (CIA) and external iliac artery (EIA) calcifications bilaterally, based on their morphology (no calcification, thin linear calcification, 1mm in thickness and bulky calcification>2mm in thickness and convex luminal margins, scores 0-3), circumference and length (no calcification, 1-25%, 26-50%, 51-75%, > 76%, scores 0-4, respectively). PCS could vary from 0-44.

Serum level of bone remodeling biomarkers will be determined on hospital admission.

Demographic and clinical data (body mass index - BMI, principal disease and additional conditions, type and duration of renal replacement therapy, KT side-and arterial segment used, hospitalization time, and graft and overall survival) will be recorded.

Patients will be followed at least one year after KT, the function of kidney transplant will be assessed by measurement of serum creatine and renal scintigraphy

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease
* operated patients (kidney transplantation)
* both gender
* older than 18 years
* written informed consent

Exclusion Criteria:

* age younger of 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo kidney transplantation in Clinical Hospital Centre Rijeka, following non-contrast CT evaluation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of iliac artery calcifications | one year
  Determination of iliac artery calcifications using CT
Distribution of iliac artery calcifications | one year
  Determination of distribution of iliac artery calcifications using CT
Determination of bone remodeling biomarker (calcium) | one year
  From the blood the bone remodeling biomarker (calcium) will be determine (mmol/l).
Determination of bone remodeling biomarker (phosphorus) | one year
  From the blood the bone remodeling biomarker (phosphorus) will be determine (mmol/l)
Determination of bone remodeling biomarker (PTH) | one year
  From the blood the bone remodeling biomarker (PTH) will be determine (pmol/l)
Determination of bone remodeling biomarker (OPG) | one year
  From the blood the bone remodeling biomarker (OPG) will be determine.
Determination of bone remodeling biomarker (RANKL) | one year
  From the blood the bone remodeling biomarker (RANKL) will be determine.
Determination of bone remodeling biomarker (GLP) | one year
  From the blood the bone remodeling biomarker (GlP) will be determine.

SECONDARY OUTCOMES:
Correlation of iliac artery calcifications with graft and overall survival in kidney transplantation patients | one year
  The investigators will found possible correlation between graft and patient survival in kidney transplantation patients
Relationship between vascular calcification burden and the serum level of bone remodeling biomarkers | One year
  The investigators will try to found correlation between vascular calcifications and serum level of bone remodeling biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Markić, Assoc.Prof., Study Chair — Clinical Hospital Center Rijeka
Locations (1):
- Clinical Hospital Center Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuza I, Dodig D, Brumini I, Tokmadzic D, Orlic L, Zgrablic D, Vukelic I, Grskovic A, Katalinic N, Jaksic A, Miletic D, Racki S, Markic D. A CT-based pelvic calcification score in kidney transplant patients is a possible predictor of graft and overall survival. Br J Radiol. 2022 Oct 1;95(1139):20220394. doi: 10.1259/bjr.20220394. Epub 2022 Oct 6. PMID 36116132
- [Background] Davis B, Marin D, Hurwitz LM, Ronald J, Ellis MJ, Ravindra KV, Collins BH, Kim CY. Application of a Novel CT-Based Iliac Artery Calcification Scoring System for Predicting Renal Transplant Outcomes. AJR Am J Roentgenol. 2016 Feb;206(2):436-41. doi: 10.2214/AJR.15.14794. PMID 26797375
- [Background] Disthabanchong S, Vipattawat K, Phakdeekitcharoen B, Kitiyakara C, Sumethkul V. Abdominal aorta and pelvic artery calcifications on plain radiographs may predict mortality in chronic kidney disease, hemodialysis and renal transplantation. Int Urol Nephrol. 2018 Feb;50(2):355-364. doi: 10.1007/s11255-017-1758-9. Epub 2017 Dec 13. PMID 29236239
- [Background] Park WY, Park SB, Han S. Long-term Clinical Outcome of Aortic Arch Calcification in Kidney Transplant Recipients. Transplant Proc. 2017 Jun;49(5):1027-1032. doi: 10.1016/j.transproceed.2017.03.072. PMID 28583520
- [Background] Benjamens S, Alghamdi SZ, Rijkse E, Te Velde-Keyzer CA, Berger SP, Moers C, de Borst MH, Slart RHJA, Dor FJMF, Minnee RC, Pol RA. Aorto-Iliac Artery Calcification and Graft Outcomes in Kidney Transplant Recipients. J Clin Med. 2021 Jan 17;10(2):325. doi: 10.3390/jcm10020325. PMID 33477285